CLINICAL TRIAL: NCT04140981
Title: Evaluation of Ultrasounographic Measurements and Anthropometric Measurements as Predictors of Difficult Direct Laryngoscopy
Brief Title: Comparison of Ultrasonographic and Anthropometric Measurements in Difficult Airway Evaluation
Status: Completed | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Kevser Peker, assitant professor, Kırıkkale University
Other Study IDs: airway ultrasounography
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Difficult Airway Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- group 1: difficult intubation according to antropometric measurements
  Interventions: Device: ultrasounography
- group 2: not difficult intubation according to antropometric measurements
  Interventions: Device: ultrasounography
- group 3: difficult intubation according to ultrasound measurements
  Interventions: Device: ultrasounography
- group 4: not difficult intubation according to ultrasound measurements
  Interventions: Device: ultrasounography

INTERVENTIONS:
Device: ultrasounography — in preoperative period, airway ultrasounagraphy for all patients will be made

SUMMARY:
In this study, anthropometric measurements (clinical measurements) will be applied in all patient groups; expected (to be difficult to provide airway patency as a result of detailed history, physical examination and evaluation tests performed by an experienced anesthesiologist), and unexpected (although it was not predicted that a difficulty was encountered). And ultrasounographic measurements will be applied in all patients. The aim of this study is to evaluate the predictive accuracy of ultrasonographic measurements.

DETAILED DESCRIPTION:
In the preoperative period, the following clinical tests will be performed before the patient arrives in the operating room and when the patient arrives, the measurements will be made by ultrasonography.

1. Mallampati classification
2. Determination of mouth opening (interinsizer distance)
3. Thyromental distance
4. Sternomental distance

Preoperative evaluation of the patients and clinical results of the airway tests (mentioned above) will be recorded. The cervical soft tissue thickness will be measured and recorded at 3 levels (thyrohyoid membrane, vocal cord, hyoid bone) with the help of ultrasonography (mentioned above). In addition, since all patients will be under general anesthesia, laryngoscopic images (laryngoscopic evaluation according to Cormack Lehane classification) routinely recorded on the anesthesia follow-up sheet will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients under general anesthesia
* ASA 1-2-3

Exclusion Criteria:

* Patients who will undergo emergency surgery,
* pregnant women,
* children,
* patients who may have difficulty in airway management due to cervical instability,
* patients with trauma or malignancy in the neck region

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ASA 1-2-3, 18-75 aged, patients undergoing general anesthesia
Sampling Method: Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Cormack Lehane classification | during the intubation period
  Laryngoscopic evaluation according to Cormack Lehane classification

SECONDARY OUTCOMES:
ultrasonographic measurement | 15 min before the operation
  Preoperative ultrasonographic measurement will be made

CONTACTS AND LOCATIONS:
Overall Officials: Kevser Peker, Principal Investigator — Kırıkkale University Faculty of Medicine
Locations (1):
- Kırıkkale Univercity Faculty of Medicine Hospital, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided